CLINICAL TRIAL: NCT01284491
Title: A Prospective, Randomized, Controlled Study to Evaluate Cutaneous Scar Quality Following Bilateral Breast Reduction With the PEAK PlasmaBlade 4.0
Brief Title: A Study to Evaluate Cutaneous Scar Quality Following Bilateral Breast Reduction With the PEAK PlasmaBlade 4.0
Acronym: PRECISE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination due to acquisition of PEAK Surgical by Medtronic
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEAK VP-00070
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Macromastia
Keywords: Breast reduction; PlasmaBlade; Electrosurgery; PEAK Surgical; Medtronic Advanced Energy; Medtronic
MeSH Terms: conditions — Gigantomastia; Hyperthermia | interventions — Electrosurgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Scalpel will be used for the skin incision and traditional electrosurgery for the subcutaneous dissection.
  Interventions: Device: Traditional Electrosurgery with scalpel
- PlasmaBlade (Experimental): The PEAK PlasmaBlade will be used for the entirety of the operation, including the skin incision.
  Interventions: Device: PEAK PlasmaBlade 4.0

INTERVENTIONS:
Device: PEAK PlasmaBlade 4.0 — The PEAK PlasmaBlade will be used for the entirety of the operation, including the skin incision.
  Other Names: PlasmaBlade
  Arms: PlasmaBlade
Device: Traditional Electrosurgery with scalpel — Scalpel will be used for the skin incision and traditional electrosurgery for the subcutaneous dissection.
  Other Names: Scalpel and electrosurgery; SOC
  Arms: Standard of Care (SOC)

SUMMARY:
The objective of this clinical study is to evaluate scar quality following incision with the PEAK PlasmaBlade 4.0 using the Patient and Observer Scar Assessment Scale (POSAS), and to compare these results to equivalently-aged scars formed following incision with a standard scalpel.

DETAILED DESCRIPTION:
Subjects attended one of two evaluation dates scheduled on January 21, 2011 and February 23, 2011. During this visit, subjects gave informed consent and were instructed on evaluating their breast reduction scars using the Patient Scar Assessment Scale. Following subjects' self-evaluation, each subject was evaluated by three evaluators using the Observer Scar Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70
2. Physically healthy, stable weight
3. Non-smokers, or prior smokers who stopped smoking at least two weeks prior to surgery.
4. Subject must understand the nature of the procedure and provide written informed consent prior to the procedure.
5. Subject must be willing and able to comply with specified follow-up evaluations.
6. Subjects who have participated in the PEAK PlasmaBlade bilateral breast reduction study.

Exclusion Criteria:

1. Age younger than 18 or greater than 70 years old
2. Anticoagulation therapy which cannot be discontinued
3. Smoking (continuous; any substance)
4. Infection (local or systemic)
5. Cognitive impairment or mental illness
6. Severe cardiopulmonary deficiencies
7. Known coagulopathy
8. Immunocompromised
9. Prior history of breast cancer
10. Kidney disease (any type)
11. Currently taking any medication known to affect healing
12. Subjects who did not participated in the PEAK PlasmaBlade bilateral breast reduction study
13. Unable to follow instructions or complete follow-up

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhay Gupta, MD, Principal Investigator — Gupta Plastic Surgery
Locations (1):
- Gupta Plastic Surgery, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects' breasts were randomized individually to the PEAK PlasmaBlade or SOC group.
Period: Overall Study
Arm/Group | Total Study Population
Started | 13
Completed | 0
Not Completed | 13
Not completed — Study termination | 13

BASELINE CHARACTERISTICS:
Arm/Group | Total Study Population
Number analyzed (Participants) | 13
Age, Customized [Number; unit: participants] — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. The protocol-specified age range is used for this baseline measure.
  participants
    18 to 70 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Scar Quality
Description: The primary endpoint will be the difference in scar quality (color, thickness, stiffness, pliability, etc.) between the scalpel and PlasmaBlade skin incisions.
Time Frame: 0-18 months following breast reduction surgery
Population: An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation.
Arm/Group | PEAK PlasmaBlade 4.0 | Traditional Electrosurgery With Scalpel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | PEAK PlasmaBlade 4.0 | Traditional Electrosurgery With Scalpel
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
Upon Medtronic's acquisition of PEAK surgical, a study integrity audit was undertaken. Results of the audit showed that patient's rights and safety were maintained, but the source data, including baseline demographics, were unverifiable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less